CLINICAL TRIAL: NCT05886556
Title: Validity of Lung Ultrasound in Diagnosis of Acute Respiratory Distress Syndrome and Prediction of Successful Weaning From Mechanical Ventilation in Those Patients
Brief Title: Validity of Lung Ultrasound in Diagnosis of Acute Respiratory Distress Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, lecture of anesthesia and surgical intensive care (Principal Investigator), Zagazig University
Other Study IDs: 8053
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: of Lung Ultrasound in Diagnosis of Acute Respiratory Distress Syndrome
Keywords: lung ultrasound, acute respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the validity of lung ultrasound compared to CT chest and chest radiograph for diagnosis of ARDS and prediction of successful weaning from mechanical ventilation in those patients compared to traditional methods.

DETAILED DESCRIPTION:
57 patients will be diagnosed as ARDS by CT chest and clinical criteria, then will be compared between the findings by lung ultrasound and chest radiograph to detect the sensitivity of both imaging to CT chest as gold standard in diagnosis of ARDS patients

ELIGIBILITY:
Inclusion Criteria:

Patients or legal guardian's consent .All patients with suspicious criteria of acute respiratory distress syndrome .Hemodynamically stable in the absence or minimal of vasopressors.

Exclusion Criteria:

Pregnant women. patients with traumatic lung injury or pneumothorax. surgical dressings over the right lower rib cage which would preclude ultrasound examination. presence of ascites. presence of lung collapse, fibrosis, or pleural effusion.

-presence of any mass or mechanical factor in the chest or the abdomen interfering with the diaphragmatic mobility.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients highly suspected to be ARDS admitted to ICU
Sampling Method: Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic data checklist | immediately after ICU admission
  Data of CT chest ,lung ultrasound and chest radiography in diagnosis of ARDS .

SECONDARY OUTCOMES:
success rate | within 24 hours after weaning
  compared the success of both methods in terms of reintubation or not for those patients
lung ultrasound as a predictor for weaning | immediately before weaning
  evaluate the scoring of lung aeration
diaphragmatic ultrasound as a predictor for weaning | immediately before weaning
  diaphragmatic thickness and excursion

CONTACTS AND LOCATIONS:
Overall Officials: mona elharisy, M.D, Study Director — zagazig university faculty of human medicine; Marwa M Medhat, M.D, Principal Investigator — zagazig university faculty of human medicine
Locations (1):
- Faculty of Medicine,Zagazig University, Zagazig, Sharqia Province, Egypt